CLINICAL TRIAL: NCT05980663
Title: Randomized Stratified Controlled Clinical Study for Evaluating the Effectiveness of a Diet Program Designed for Reducing Body Weight Using Standard and Innovative Products in Obese Participants With Asthma
Brief Title: Evaluation of the Effectiveness of Standard and Innovative Products That Represent a Substitute Meal for Weight Management in a Reduction Diet in Obese Participants With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital Srebrnjak (Other)
Collaborators: Belupo (Other); Podravka d.d. (Unknown)
Responsible Party: Principal Investigator, Mirjana Turkalj, MD, Professor, MD, PhD, Children's Hospital Srebrnjak
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KK.01.1.1.07.0075_2
Record Dates: First submitted 2023-05-22; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Asthma; Overweight
Keywords: obesity; asthma; overweight; nutrition
MeSH Terms: conditions — Obesity; Asthma; Overweight

STUDY DESIGN:
Intervention Model Description: Randomized stratified controlled clinical study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active group (Experimental): Participants use the innovative line of products intended for body weight reduction, that represent a meal replacement for weight management.
  Interventions: Dietary Supplement: Meal replacement product- INNOVATIVE PRODUCT
- Active control (Active Comparator): Participants use the standard line of products intended for weight reduction that represent a meal replacement for weight management with already proven clinical effectiveness (positive control).
  Interventions: Dietary Supplement: Meal replacement product- STANDARD PRODUCT
- Control group (No Intervention): Participants receive personalized advice on proper nutrition for a reduction diet in which they use common food.

INTERVENTIONS:
Dietary Supplement: Meal replacement product- STANDARD PRODUCT — standard product line contains common ingredients and this type of product already exists on world markets
  Arms: Active control
Dietary Supplement: Meal replacement product- INNOVATIVE PRODUCT — innovative product line contains raw materials that are considered better sources of potentially bioactive components
  Arms: Active group

SUMMARY:
Randomized stratified controlled clinical study for evaluate the effectiveness of a diet program designed for reduce body weight through standard and innovative products that are a substitute meal for weight management in a reduction diet in obese participants with asthma.

DETAILED DESCRIPTION:
In the last few decades, there has been an increase in the number of obese people to the level of a global epidemic as a result of inadequate diet, sedentary lifestyle, but also genetic predispositions. The World Health Organization (WHO) declared obesity to be the biggest, global, chronic health problem in adults, that is increasingly becoming a more serious problem than malnutrition.On the other hand, obesity is a risk factor for the development of contemporary non-infectious diseases today that account for more than 80% of mortality in developed countries, such as vascular disease, diabetes and respiratory diseases such as asthma.

This trend is also recorded in Croatia, both in adult population and in children if the data from 2003 and 2015 are being compared, while according to data from 2019, almost two thirds of the adult population in Croatia were overweight or obese (42% overweight, 23% obese).

Of particular concern are the data from the European Obesity Monitoring Initiative from 2018/2019. according to which in Croatia 35% of children aged 8.0 to 8.9 were overweight or obese. At the national level, the problem of obesity is greater in boys than in girls, and it is 17.8% compared to 11.9% of girls. Croatia is in a high fifth place together with other countries of the Mediterranean region of Europe due to the shift from the Mediterranean to the Western lifestyle.

In cooperation with Podravka, Belupo has developed a standard and innovative product line. Products are replacing one or more one or more daily meals, and thay must comply with Regulation 2016/1413 requirements related to energy value, content and composition of fats and proteins, the amount of vitamins and minerals in this type of products.

The standard product line contains common ingredients and this type of product already exists on world markets, while the innovative product line differs from the standard one by implementing raw materials that are considered better sources of potentially bioactive components.

The study for a group of adult participants was designed in such a way that the participants in the initial stage follow a low-calorie diet of about 1000 - 1100 kcal, whereby 5 daily meals are replaced with meal replacements in the reduction diet (active group and active control) (intensive phase). In subsequent stages, subjects gradually increase their energy intake and gradually substitute meal replacement product (MRP) with regular nutritionally profiled meals (active phase and maintenance phase). The final (stable) phase represents the stage in which, in addition to one meal replacement per day, the usual meals designed by the nutritionists of Belupo and the Culinary Center of Podravka are consumed, where education and nutrition counseling is also carried out.

The study for the child population of respondents is designed in such a way that the respondents in the initial phase implement a low-calorie diet of about 1300-1500 kcal, whereby 3 daily meals are replaced with meal replacements in the reduction diet in addition to 2 nutritionally balanced regular meals that include a minimum of 5 daily servings of fruits and vegetables (active group and active control) (intensive phase).

In subsequent phases, subjects gradually increase their energy intake and gradually replace MRP with regular nutritionally profiled meals (active phase and stable phase). The final phase represents the phase in which subjects consume the usual meals designed by the nutritionists of Children's hospital Srebrnjak, where education and nutrition counseling is also carried out.

The usual meals of the later stages of the study, apart from being low in energy and highly nutritionally dense are composed in such a way that they are either ready for consumption as a complete meal (e.g. ready- to eat tuna salad) or can be quickly prepared. In this way, the test respondents are directed to an adequate diet, which, by adopting proper food and lifestyle habits, will ultimately enable them to maintain the achieved reduced body weight in the long term.

Study entry stage (0-2 weeks): subjects are recruited respecting the inclusion and exclusion criteria. Recruitment is carried out by a doctor. During this stage, subjects replace standard meals with meal replacement products and reduce energy intake to a final defined intake depending on the group of subjects.

200 participants in a ratio of 2:1:1 (adults and children)

* active group - 80
* active control (positive control group) - 80
* control group (negative control group) - 40

Adult participants program:

The daily energy intake is defined at around 1000-1100 kcal per day, and counseling on nutrition and physical activity is carried out.

1. Intensive phase(2-14 weeks) about 1000 - 1100 kcal/day 5 MRP (200-220 kcal per product) + 1 salad (20 kcal per portion) + water/unsweetened tea.
2. Active phase(14-21 weeks) 1100-1200 kcal/day 3 MRP (200-220 kcal per meal) + 2 regular meals (200-280 kcal) + water/unsweetened tea.
3. Maintenance phase (21-28 weeks): 1200-1500 kcal/day 2 MRP (200-220 kcal per meal) + 3 regular meals (260-350 kcal) + water/unsweetened tea
4. Stable phase (28-40 weeks): 1500-2000 kcal 1 MRP (200-220 kcal per meal) + 4 regular meals (approx. 320-450 kcal) + water/unsweetened tea Usual meals can also contain snacks with lower energy values, but it is important to consume approx. 1300-1800 kcal per day with usual foods.

Children participants program:

The daily energy intake is defined at around 1300-1500 kcal per day, and counseling on nutrition and physical activity is carried out.

1. Intensive phase children (weeks 2-14) around 1300-1500 kcal/day 3 MPR (200-220 kcal per product + 2 regular meals (320-400 kcal) + 1 or more salad (20 kcal per product)+ water/unsweetened tea.
2. Active phase children (14-21 weeks) around 140-1600kcal/day 2 MPR (200-220 kcal per product) + 3 regular meals (320-400 kcal) + water/unsweetened tea.
3. Maintenance phase (21-28 weeks): 1600-1900 kcal/day 1 MRP (200-220 kcal per meal) + 4 regular meals (350-420 kcal) + water/unsweetened tea
4. Stable phase children (week 28-40) 1750-2250 kcal/day. 5 regular meals (350-450 kcal) + water/unsweetened tea.

Snacks are included in regular meals, where the total value of meals and snacks does not exceed the total set value of regular meals.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-60, children aged 12-18
* both sexes
* BMI >27 kg/m2 (adults); > 90th centile for BMI (children)
* clinical diagnosis of asthma
* signed informed consent

Exclusion Criteria:

* significant comorbidities: uncontrolled diabetes mellitus requiring insulin therapy and other endocrine disorders, cardiovascular disorders and other chronic diseases (including malignancies), chronic inflammatory diseases of the gastrointestinal tract, mental disorder
* people who are currently on or have recently gone through a weight loss program (in the past 3 months)
* people who in the past 6 months had an unwanted and uncontrolled loss of body weight >5%
* people who underwent bariatric surgery in the past 6 months.
* people using drugs that increase or decrease appetite
* permanent therapy with steroid drugs, antidepressants, cytostatics, hormone therapy, beta-blockers, etc.
* people with eating disorders (bulimia)
* alcohol and drug addicts
* pregnancy, breastfeeding
* unstable thyroid disease

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
BM/FM | every 4 weeks, through study completition (up to 9 months)
  To determine the effectiveness of a weight change diet program based on an innovative and standard product line through actual reduction of the body mass (BM) / fat mass (FM) of the participants in relation to their pre - trial body mass(BM)/fat mass (FM).

SECONDARY OUTCOMES:
Anthropometric measurements | every 2 months, through study completition (up to 9 months)
  Change in anthropometric measurements- waist and hip circumference and waist/hip ratio and waist/height ratio
  Measurements of participants' waist, hip and height in meters will be taken. This multiple measurements will be aggregated and presented in ratio waist [meter] / hip [meter] and ratio waist [meter] / height [meter]
Lipid profile (triglycerides, total cholesterol, HDL, LDL) | at 1st week of the study and after 3, 6 and 9 months, through study completition (up to 9 months)
  Change of the cholesterol test/lipid panel/lipid profile (change in HDL/LDL ratio) compared to initial values
Questionnaire on quality of life | at the beginning of the study (1st week) and at the end (40th week)
  The questionnaire consists of descriptive system and visual analogue scale.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The visual analogue scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
  The questionnaire is in Croatian language, with a valid and accurate translation of the corresponding original document.
Change of asthma control | every 3 months, through study completition (up to 9 months)
  ACT Questionnaire will be used to tell us if the asthma treatment plan is optimal and if asthma is being properly controlled. Maximal score is 25, where higher scores reflect greater asthma control while if the score is 19 or less that may be a sign that asthma is not controlled as well as it could be.
Change in the number of asthma exacerbations and severity | every 3 months,through study completition (up to 9 months)
  The the number of exacerbations will be recorded along with the therapy used (use of salbutamol, oral or parenteral corticosteroids etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, Croatia